CLINICAL TRIAL: NCT06048276
Title: Miscarriage Preventing Herbal Medicines and the Risk of Birth Defects: a Population-based Cohort Study
Status: Active, not recruiting | Type: Observational
Sponsor: West China Hospital (Other)
Collaborators: Xiamen Health Commission (Unknown); Xiamen Health and Medical Big Data Center (Unknown)
Responsible Party: Principal Investigator, Sun Xin, Director of Chinese Evidence-based Medicine Center, West China Hospital
Other Study IDs: HERB and BD
Record Dates: First submitted 2023-09-14; First posted 2023-09-21 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Pregnancy; Birth Defects; Drug Exposures
Keywords: Herbal medicines; Birth defects; Drug exposures; Cohort study
MeSH Terms: conditions — Congenital Abnormalities | interventions — Plant Extracts

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Drug exposure: Herbal medicines
  Interventions: Drug: Herbal medicines (e.g., Yunkang granules, Duzhong granules)

INTERVENTIONS:
Drug: Herbal medicines (e.g., Yunkang granules, Duzhong granules) — Herbal medicines (e.g., Yunkang granules, Duzhong granules) exposure at the early gestation.

SUMMARY:
Using data from a population-based medicine use cohort in Xiamen, China, this retrospective cohort study will investigate whether herbal medicines used to prevent miscarriage are associated with increased risk of birth defects.

DETAILED DESCRIPTION:
Herbal medicines have a long history of use for pregnant women both in China and around the world. However, the safety of herbal medicines used at the early gestation is often questioned regarding their impact on offspring. Therefore, the aim of this study is to investigate whether miscarriage preventing herbal medicines associated with increased risk of birth defects.

A large medication use cohort will be developed by linking a population-based pregnancy registry (i.e., REPRESENT) and a population-based pharmacy database, which documented all prescriptions at both outpatients and inpatients from conception to delivery. This cohort will include herbal medicines formula which were granted approval by the Chinese National Medical Products Administration.

Using data from this cohort, the investigators will investigate the prevalence of the use of herbal medicine formulas and prescription patterns at the first trimester. This study will then investigate the association between miscarriage preventing herbal medicines and the risk of birth defects. A propensity score matching (PSM) based Poisson regression will be used to estimate the relative risk. To ensure the robustness of the results investigators will perform several sensitivity analyses and negative control analyses, such as restricting the population to women with singleton pregnancies, excluding individuals who had undergone in vitro fertilization (IVF), and considering those women who were prescribed herbal medicines during the middle and late stages of pregnancy as the negative exposure control group.

ELIGIBILITY:
Inclusion Criteria:

* Pregnancies registered at REPRESENT and underwent live births between January 2013 and December 2018 were included.

Exclusion Criteria:

* (1) those with the first antenatal visit occurring after 20 gestational weeks, (2) those without timing records of the last menstrual period or delivery dates, (3) those with known factors related to birth defects (e.g.,syphilis positive, epilepsy), (4) those prescribed known medications associated with birth defects (e.g.,dezocine, diazepam).

Ages: 15 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — All pregnant women registered at the REPRESENT were enrolled.
Study Population: Between January 2013 and December 2018, all pregnant women who registered at the REPRESENT in Xiamen was included in this cohort.
Sampling Method: Probability Sample
Enrollment: 200000 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-10-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall birth defects (excluding chromosomal malformations) | From conception to 42 days after delivery
  Number of births with birth defects

SECONDARY OUTCOMES:
National monitored 23 main types of birth defects | From conception to 42 days after delivery
  Number of births with 23 major births defects defined by National Health Standard Criteria in the China national universal surveillance system

CONTACTS AND LOCATIONS:
Overall Officials: Xin Sun, PHD, Study Chair — Chinese Evidence-based Medicine Center, West China Hospital, Sichuan
Locations (1):
- Xiamen Health and Medical Big Data Center, Xiamen, Fujian, China

IPD SHARING:
Plan to Share IPD: Yes
Following the policy of Xiamen Health Commission, research institutions could apply for data access by submitting a formal study protocol, subjected to approval by the Xiamen Health and Medical Big Data Center and the Chinese Evidence-based Medicine Center. Ethical review and research registration are mandatory for all studies.
Supporting Information: Study Protocol, SAP